CLINICAL TRIAL: NCT06203964
Title: Organizing Pneumonia in Lung Transplant Recipients, a Restrospective Exploratory Study (OPIL-Study)
Acronym: OPIL
Status: Active, not recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00824
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Organizing Pneumonia; Lung Transplant Rejection
MeSH Terms: conditions — Organizing Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The aim of this study is to generate evidence regarding organizing pneumonia in lung transplant recipients.

DETAILED DESCRIPTION:
Allograft failure remains the leading cause of morbidity and mortality in lung transplant recipients (LTR) accounting for 40% of deaths beyond the first year after transplantation. The current median survival over all LTRs is 6.0 years. Chronic allograft dysfunction (CLAD) is defined as a substantial and persistent decline in the measured forced expiratory volume in 1 second (FEV1) with ≥ 20% from the baseline value. The consensus statement from the International Society for Heart and Lung Transplantation in 2019 classified CLAD into two main phenotypes: Bronchiolitis obliterans syndrome (BOS) and restrictive allograft syndrome (RAS). Based on respiratory function and computed tomography (CT) findings, CLAD is classified into four groups: BOS, RAS, mixed (BOS and RAS), and undefined. Definite CLAD-BOS is defined as persistent decline of ≥ 20% from the reference value after more than 3 months without a restriction and without persistent radiologic pulmonary opacities.

The main histologic findings of BOS include obliterative bronchiolitis (OB) accompanying chronic inflammation and fibrosis in the respiratory tract.

Up to 30 % of patients with CLAD present a restrictive pattern stated as CLAD-RAS. CLAD-RAS is physiologically defined as a persistent decline in FEV1 (± FVC) of ≥20% compared with the reference or baseline value, a decrease in total lung capacity (TLC) to ≤90% compared with baseline and the presence of persistent opacities on chest imaging. The pathology of RAS is nearly identical to that observed in the entity of pleuroparenchymal fibroelastosis. It features severe alveolar fibrosis organized around the pleura and the interlobular septa with concomitant obliterative bronchiolitis lesions. Von der Thüsen et al. analysed tissue samples of 21 patients with RAS describing not only patterns consistent with pleuroparenchymal fibroelastosis but also nonspecific interstitial pneumonia, irregular emphysema, organizing pneumonia (OP) and acute fibrinous organizing pneumonia (AFOP).

Some authors have advocated acute fibrinoid and organizing pneumonia (AFOP) as a third potential form of chronic allograft dysfunction, with decline of lung functions as for CLAD but with distinct histopathology and imaging findings. Paraskeva et al. identified AFOP as a novel entity in 22 out of 194 (11%) lung transplant recipients, invariably associated with a rapid decline in respiratory function and death after a median time of 101 days. AFOP is a unique pathological entity with intra-alveolar fibrin in the form of "fibrin balls" and organizing pneumonia.

While AFOP and its clinical impact is getting more and more recognized as a pattern of RAS, little is known about OP and its clinical impact in LTRs. OP per se is a pattern of lung tissue repair after injury. It can be a response to a specific lung injury (secondary OP) or cryptogenic (COP). COP has no identifiable cause and is classified as a form of idiopathic diffuse parenchymal lung disease (DPLD). So far it is not clear if OP is a form of the RAS spectrum and if the presence of OP might also predict a rapid decline in lung function and survival comparable with AFOP.

The aim of this study is to investigate the prevalence of OP forms in lung transplant recipients, possible risk factors for OP and the impact of OP itself on the course of lung allograft function.

ELIGIBILITY:
Inclusion Criteria:

* All lung transplant recipients treated in the lung transplantation department of the USZ will be included in this analysis with documented tissue sampling or autopsy between 01.01.2012 and 01.06.2023

Exclusion Criteria:

* Denied general consent or any statement verbal or in writing by patient that precludes research

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All lung transplant recipients treated in the lung transplantation department of the USZ will be included in this analysis with documented tissue sampling or autopsy between 01.01.2012 and 01.06.2023
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2023-07-07 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of organizing pneumonia | 01.01.2012-01.06.2023

SECONDARY OUTCOMES:
Body Mass Index | date of organizing pneumonia
Forced expiratory volume in 1 second | 1 year before and after organizing pneumonia
Total lung capacity | 1 year before and after organizing pneumonia
Vital capacity | 1 year before and after organizing pneumonia
Prevalence of primary graft dysfunction | 01.01.2012-01.06.2023
Cell count of eosinophils in blood | 1 year before and after organizing pneumonia
Cell count of lymphocytes in blood | 1 year before and after organizing pneumonia
Cell count of neutrophils in blood | 1 year before and after organizing pneumonia
Level of rhematoid factor in blood | date of organizing pneumonia
Level of anti-nuclear antibodies in blood | date of organizing pneumonia
Level of antineutrophil cytoplasmic antibodies in blood | date of organizing pneumonia
Prevalence of infection | date of organizing pneumonia
C-reactive proteine | date of organizing pneumonia
Histopathological patterns beside organising pneumonia | date of organizing pneumonia
Radiological findings in CT scan | date of organizing pneumonia
Medication associated with organizing pneumonia | date of organizing pneumonia
NTproBNP | date of organizing pneumonia
Echocardiography | 1 year before and after organizing pneumonia
Cellcount in the bronchoalveolar lavage | 1 year before and after organizing pneumonia
Level of donor specific antibodies | 1 year before and after organizing pneumonia
Time to death | after diagnosis of organizing pneumonia
Reason for death according to biopsy results od physician declared cause of death | after diagnosis of organizing pneumonia (- 01.06.2023)
Number of patients with therapeutic interventions due to organizing pneumonia | 01.01.2012-01.06.2023
Prevalence of risk factors of OP | 01.01.2012-01.06.2023
  * Prevalence of infection (Virus/Bacteria/Fungus)
  * CMV/EBV PCR results
  * Graft ischemic time
  * Prevalence and type of malignant diseases (eg PTLD)
  * Rheumatic disease (Connective tissue disease, vasculitis)
  * GERD with aspiration (upper endoscopy findings or pH-metric findings)
  * Common variable immunodeficiency
  * Inflammatory bowel syndrome
  * Medication or monitoring non-compliance
  * Radiation
  * Malignant disease

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided